CLINICAL TRIAL: NCT04395040
Title: Identify the Obstacles to Early Diagnosis of Cancer in Patients Over 75 Years Old, on an Outpatient Basis
Acronym: DPCMG
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0731
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Cancer; Aging
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Elderly patients with digestive cancer or breast cancer.
  Interventions: Other: Semi-structured interview

INTERVENTIONS:
Other: Semi-structured interview — Semi-structured interview

SUMMARY:
A third of cancers are diagnosed in patients over 75 years of age. There are fears of the elderly talking about new symptoms. The doctor may find himself trapped by general symptoms, which can be confused with "normal aging".

Some older, younger people have lived in a world where cancer was little talked about, where there was little treatment possible.

There is an idea that doctors are not very quick to start curative treatment because they think that the elderly cannot bear it.

It is important to differentiate screening and early diagnosis.

Delayed treatment causes a decrease in survival and quality of life. Cancer can be discovered suddenly: for example, occlusion with peritonitis in case of a stenosing colonic tumor, leading to urgent management.

The elderly are often excluded from clinical studies.

In addition, the geriatric population is heterogeneous, leading to very diverse and individual care, with prioritization of issues.

Oncogeriatrics, which combines two services (oncology and geriatrics), is a specialized discipline, promoting comprehensive care for the elderly patient with cancer.

The general practitioner is at the center of care. It detects early signs and starts examinations if necessary.

Cancer care can be divided up with the different stages of care with various teams, including organ specialists.

The general practitioner is the privileged interlocutor for the patient and their family (medico-psycho-social plan), who knows their history and their experience.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 75 years old (terminal included)
* Incident diagnosis
* Has cancer whose diagnosis dates back more than 3 months
* Digestive cancer, breast cancer
* Stage of advanced cancer (TNM stage: T> T2 (terminal included), M1)
* According to the opinion of the oncogeriatrician on the time of taking charge
* Follow-up of a geriatrics service, onco-geriatrics orientation
* Living in the Rhône department
* Non-opposition of the patient to the study

Exclusion Criteria:

* Cancer diagnosis more than 6 months old
* Patient denies

Min Age: 75 Years | Sex: All
Age Groups: Older Adult
Study Population: Elderly patients with digestive or breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-02 (Actual)

PRIMARY OUTCOMES:
Identify the obstacles to the early diagnosis of cancer in patients over 75 years old suffering from cancer. | 1 hour
  Explore, during a semi-structured interview with the patient, the brakes and levers:
  * related to the patient
  * linked to the doctor: felt on the practices of health professionals, paternalistic, patient-centered approach
  * linked to the disease: symptoms, acceptance of examinations, acceptance of diagnosis
  * linked to society

CONTACTS AND LOCATIONS:
Overall Officials: Camille TAZELMATI, MD Student, Principal Investigator — Hospices Civils de Lyon; Marie VALERO, MD, Study Director — Hospices Civils de Lyon
Locations (3):
- France (3):
  - Centre Léon Bérard, Lyon
  - Hôpital Lyon Sud, Pierre-Bénite
  - Centre hospitalier Fleyriat, Viriat